CLINICAL TRIAL: NCT06578325
Title: Effects of Thai Dance Meditation Exercise on Renal and Cerebrovascular Function in Elderly With Diabetic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Prof. Dr.Daroonwan Suksom, Faculty of Sports science, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPSC-9
Record Dates: First submitted 2024-08-18; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Diabetic Kidney Disease
Keywords: Diabetic kidney disease; Cerebrovascular reactivity; Renal function; Thai dance meditation
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes kidney disease patients with Thai dance meditation (Experimental): Male and female diabetic kidney disease patients were selected based on screening for diabetes and renal function. They were recruited for measurement of all variables in the study to compare with another group.
  Interventions: Other: Thai dance meditation
- Diabetes kidney disease patients (Sham Comparator): Male and female diabetic kidney disease patients were not training Thai dance meditation. They were recruited for measurement of all variables in the study to compare with another group.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Thai dance meditation — Thai dance meditation training program will be based on aerobic Thai dance exercise combined with Buddhist meditation. The participants will perform aerobic Thai dance meditation while concentrated on hand movements through counting the numbers 1 2 3 4 5 6 7 1 on the 1st round and continuing on the 2nd round, counting as 1 2 3 4 5 6 7 2…. Repeat for 8 rounds. Thai dance meditation will be conducted at mild to moderate intensity (40-60% heart rate reserve) and in phase 2 (week 7-12), the training intensity will be increased to moderate intensity (50-60% heart rate reserve). In both phases the training will be performed foe 50 minutes, 3 times per week.
  Arms: Diabetes kidney disease patients with Thai dance meditation
Other: No intervention — No intervention
  Arms: Diabetes kidney disease patients

SUMMARY:
Elderly with diabetic kidney disease who practiced Thai dance meditation training more favorable adaptations than normal daily life in improving glycemic control, kidney function, vascular function and cerebrovascular function.

DETAILED DESCRIPTION:
This cross-sectional study was to compare glycemic control, kidney function, vascular function, cerebrovascular function, physical fitness and quality of life between elderly with diabetic kidney disease who practiced Thai dance meditation training and normal daily life.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria included diabetic kidney disease (DKD) (as defined by the KDIGO (Kidney Disease Improving Global Outcomes 2012), a baseline glycosylated hemoglobin (HbA1c) value of 7-9%, albumin-to creatinine ratio (ACR): A3 [>300 mg/day; ACR, >300 mg/g (>30 mg/mmol)], GFR category 3 (moderately decreased) has now been divided into categories G3a [45-59 mL/ min1 /(1.73m2) and G3b [30 -44 mL/ min1/(1.73 m2) which represent mildly to moderately decreased function and moderately to severely decreased function and no previous exercise training in the past 6 months.
* All participants were free from diabetic retinopathy, severe diabetic neurophathy, severe cardiovascular and cerebrovascular diseases.
* Participants had Montreal Cognitive Assessment - Thai (MoCa-T) scores between 18 24 points.
* Not having uncontrolled high blood pressure (Systolic blood pressure; SBP) >159 mmHg and Diastolic blood pressure; DBP) > 99 mmHg

Exclusion Criteria:

- Participants were excluded if they dropped out or completed less than 80% of the training schedule

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Change from baseline systolic blood pressure, diastolic blood pressure, and mean arterial pressure at 12 weeks.]
  Blood pressure (systolic blood pressure, diastolic blood pressure, and mean arterial pressure) in mmHg will be measured with automated blood pressure in mmHg device (CARESCAPE V100, GE Dinamap).
Heart rate | Change from baseline heart rate at 12 weeks
  Heart rate in beats per minute will be measured with automated blood pressure in beat per minute device (CARESCAPE V100, GE Dina map).
Body fat | Change from baseline body fat at 12 weeks
  Body fat in percent will be measured with dual energy x-ray absorptiometry in percent (Prodigy-Pro, GE healthcare).
Muscle mass and Weight | Change from baseline muscle mass and weight at 12 weeks.
  Muscle mass and weight in kilograms will be measured with dual energy x-ray absorptiometry in kilogram (Prodigy-Pro, GE healthcare).
Arterial stiffness | Change from baseline brachial-ankle pulse wave velocity at 12 weeks
  Arterial stiffness will be measured with brachial-ankle pulse wave velocity in centimeter per second (VP-1000 plus, omrom Healthcare).
Macro vascular function | Change from baseline brachial artery flow-mediated dilatation at 12 weeks
  Macro vascular function will be measured by brachial artery flow-mediated dilatation in percent with ultrasonography equipment EPIQ 5G, Phillips.
Renal function | Change from baseline Blood urea nitrogen at 12 weeks.
  Blood urea nitrogen (BUN) in milligram per deciliter will be measure by Kinetic test with urease and glutamate dehydrogenase with urease/glutamate dehydrogenase coupled enzymatic (Coupled enzymes)
Intrarenal artery | Change from baseline renal arterial resistive index (RI) at 12 weeks.
  Intrarenal artery will be measured by renal blood flow in renal arterial resistive index (RI) with ultrasonography equipment EPIQ 5G, Phillips.
Post Occlusive Reactive Hyperemia; PORH | Change from baseline Post Occlusive Reactive Hyperemia; PORH at 12 weeks.
  Evaluation of blood flow to the skin area in percent will be measured by Post Occlusive Reactive Hyperemia in percent; PORH with Laser Doppler flowmeter, Perimed AB, Sweden.
Cerebral blood flow | Change from baseline cerebral blood flow at 12 weeks
  Cerebral blood flow in centimeter per second will be measure with ultrasonography equipment (EPIQ 5G, Phillips).
Cerebrovascular conductance index | Change from baseline cerebrovascular conductance index at 12 weeks
  Cerebrovascular conductance index in cm/sec/mmHg will be measured with ultrasonography equipment (EPIQ 5G, Phillips).
Cerebrovascular reactivity index | Change from baseline cerebrovascular reactivity index at 12 weeks
  Cerebrovascular reactivity index in %cm/sec/mmHg will be measured with ultrasonography equipment (EPIQ 5G, Phillips).
Arterial compliance | Change from baseline Arterial compliance at 12 weeks
  Arterial compliance in units will be measure by carotid diameter during systolic and diastolic with ultrasonography equipment (EPIQ 5G, Phillips) and systemic blood pressure with (VP-1000 plus, omrom Healthcare).
Pulsatility index | Change from baseline Pulsatility index at 12 weeks.] 12.Montreal Cognitive Assessment
  Pulsatility index in units will be measure with ultrasonography equipment (EPIQ 5G, Phillips).
Montreal Cognitive Assessment | Change from baseline Montreal Cognitive Assessment at 12 weeks.]
  Montreal Cognitive Assessment in score (0 - 30 scores) cut off below 25 scores that indicate impairment cognitive function.
Mini-Mental State Examination | Change from baseline Mini-Mental State Examination at 12 weeks.]
  Mini-Mental State Examination in scores (0 - 30 scores) cut off below 25 scores that indicate impairment cognitive function.
Trail Making Test-B | Change from baseline Trail Making Test-B at 12 weeks
  Trail Making Test-B in second cut off below 101 seconds that indicate dementia.
Fasting blood sugar | Change from baseline fasting blood sugar at 12 weeks.]
  Fasting blood sugar in mg/dl will be measure with enzymatic assay using hexokinase reaction.
Glycosylated hemoglobin | Change from baseline Glycosylated hemoglobin at 12 weeks.]
  Glycosylated hemoglobin in percent will be measure with enzymatic assay using hexokinase reaction.
Homeostasis Model Assessment of insulin resistance | Change from baseline Homeostasis Model Assessment of insulin resistance at 12 weeks.]
  Homeostasis Model Assessment of insulin resistance in units will be calculated with Fasting blood sugar and insulin.
Creatinine | Change from baseline creatinine at 12 weeks.]
  Creatinine in mg/dl will be measure with enzymatic assay
estimate Glomerular filtration rate | Change from baseline estimate Glomerular filtration rate at 12 weeks.]
  estimate Glomerular filtration rate in ml/min/1.73 m2 will be calculated by CKD-EPI formular according to National kidney foundation recommendation.
Cystatin C | Change from baseline blood urea nitrogen at 12 weeks
  Cystatin C in mg/L will be measure with particle enhanced Immunoturbidimetric assay
Urine albumin creatinine ratio | Change from baseline urine albumin creatinine ratio at 12 weeks.
  Urine albumin creatinine ratio will be measure with Immunoturbidimetric assay
Stroop test | Change from baseline Stroop test in second at 12 weeks.
  Stroop test in second will be measured with EncephalApp - Stroop Test

SECONDARY OUTCOMES:
Waist circumference | Change from baseline waist circumference at 12 weeks]
  Waist circumference in inch will be measure by waist tape
.Flexibility testing | Change from baseline Chair sit & reach at 12 weeks.]
  Flexibility testing will be measure by Chair sit & reach protocol in centimeters.
Muscle strength testing | Change from baseline arm-curl and chair stand at 12 weeks.]
  Muscle strength testing will be measured by arm-curl test repetitions in 30 seconds
Muscle strength testing | Change from baseline arm-curl and chair stand at 12 weeks.]
  Muscle strength testing will be measured by arm-curl test and chair stand test in repetitions in 30 seconds
Balance testing | Change from baseline time up and go at 12 weeks.]
  Balance testing will be measured by time up and go testing in seconds.
Cardiopulmonary fitness | Change from baseline 6-minutes walk at 12 weeks.]
  Cardiopulmonary fitness will be measure by 6-minutes walk test in meters.
Lipid profile | Change from baseline Nitric oxide at 12 weeks.] cholesterol, triglyceride, high density lipoprotein, and low density lipoprotein at 12 weeks.]
  Lipid profile will be measure by cholesterol, triglyceride, high density lipoprotein, and low density lipoprotein in mg/dl.
Interleukin-6 (IL-6), Tumor necrosis factor-alpha (TNF- α), Brain derived neurotrophic factor, Malondialdehyde, Superoxide Dismutase. | Change from baselineInterleukin-6 (IL-6), Tumor necrosis factor-alpha (TNF- α), Brain derived neurotrophic factor, Malondialdehyde, Superoxide Dismutase. at 12 weeks.]
  Interleukin-6 (IL-6), Tumor necrosis factor-alpha (TNF- α), Brain derived neurotrophic factor, Malondialdehyde, Superoxide Dismutase in pg/ml will be measure with ELISA assay kit.
Nitric oxide | Change from baseline Nitric oxide at 12 weeks.
  Nitric oxide in µM will measured with standard Griess reagents.
Quality of life in patients with chronic kidney disease | Change from baseline at 12 weeks.
  Quality of life will be measured by SF-36 questionnaire for evaluation of Quality of Life in patients with chronic kidney disease. The scores of questionnaires were 75-100 points for good quality of life, 50-75 points for moderate quality of life, 25-50 points for low quality of life and 0-25 points for very low quality of life.
Flexibility testing | Change from baseline back scratch at 12 weeks.
  Flexibility testing will be measure by back scratch in centimeters.
Muscle strength testing | Change from baseline chair stand at 12 weeks.]
  Muscle strength testing will be measured by chair stand test in repetitions in 30 seconds
Body mass index (BMI) | Change from baseline BMI at 12 weeks.
  Body mass index (BMI) through height and weight measurement by body composition analyzer weight and height will be combined to report BMI in kg/m^2.

CONTACTS AND LOCATIONS:
Overall Officials: Daroonwan Suksom, Ph.D., Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Sports Science, Chulalongkorn University, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No